CLINICAL TRIAL: NCT05255328
Title: Clinical Long Term Evaluation of Glutamine Supplement in MELAS (Mitochondrial Encephalopathy, Lactic Acidosis, and Stroke-like Episodes) Syndrome in Order to Prevent Neurological Damage.
Brief Title: Clinical Long Term Evaluation of Glutamine Supplement in MELAS Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Jesús González de la Aleja Tejera, Jesús González de la Aleja Tejera, MD, PhD, Principal Investigator, Hospital Universitario 12 de Octubre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLN-9-MIT2
Record Dates: First submitted 2022-01-19; First posted 2022-02-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: MELAS Syndrome
Keywords: MELAS; Glutamine; Oral supplements; Amino acids
MeSH Terms: conditions — MELAS Syndrome

STUDY DESIGN:
Intervention Model Description: Glutamine oral supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MELAS (Experimental): Patients with MELAS syndrome will receive 12-18g/day of glutamine
  Interventions: Dietary Supplement: Glutamine oral supplement

INTERVENTIONS:
Dietary Supplement: Glutamine oral supplement — 12-18 g /day of glutamine supplementation

SUMMARY:
The purpose of this study is to assesses the clinical efficacy of oral supplementation with glutamine over 3 years.

DETAILED DESCRIPTION:
Mitochondrial encephalomyopathy, lactic acidosis, and stroke-like episodes (MELAS) syndrome is a genetically heterogeneous disorder. The most common mutation is in the mtDNA gene MT-TL1 encoding the mitochondrial tRNALeu (UUR). For understanding the development of seizures in patients with mitochondrial disease, a study has recently emphasized the deficiency of astrocytic glutamine synthetase, creating a disinhibited neuronal network for seizure generation. The investigators propose to evaluate nine patients with mitochondrial DNA mutation and MELAS. Patients will receive oral supplementation with 12-18 g/day of glutamine (adjusted for weight and plasma concentrations). The primary outcome measures modification in clinical scales.

ELIGIBILITY:
Inclusion Criteria:

* MELAS syndrome Clinically and genetically confirmed.
* Patients have already participated in GLN-9-MIT study

Exclusion Criteria:

* subjects harboring a MELAS-related pathogenic mtDNA mutation no fulfilling the complete diagnostic criteria for the MELAS phenotype

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2024-07-24 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy; JMDRS | 36 months
  Change from Baseline clinical scale (Japanese mitochondrial disease rating scale (JMDRS)) at 12,24,36 months to test Clinical efficacy of oral supplementation
Clinical efficacy; MMSE | 36 months
  Change from Baseline cognitive test (Mini-Mental State Examination (MMSE)) at 12,24,36 months to test Clinical efficacy of oral supplementation

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 36 months
  To recorde all adverse events grades; with special interest on investigations (CTCAE v5.0, 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Jesús González de la Ajeja Tejera, MD, PhD, Principal Investigator — Hospital Universitario 12 Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain